CLINICAL TRIAL: NCT04296786
Title: Sintilimab Combined With Chidamide in the Treatment of Relapsed and Refractory Cutaneous T-cell Lymphoma: a Multicenter Single Arm Phase II Study
Brief Title: Sintilimab Plus Chidamide in the Treatment of Relapsed and Refractory Cutaneous T-cell Lymphoma: a Multicenter Phase II Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Peking University Third Hospital (Other); Beijing Longfu Hospital (Unknown); Dongzhimen Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-NHL-006
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-01

CONDITIONS: Cutaneous T-cell Lymphoma
Keywords: Chidamide; Sintilimab; cutaneous T-cell lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous | interventions — sintilimab; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chidamide plus Sintilimab (Experimental): Patients in experimental group will receive fixed does of Sintilimab and Chidamide. This regimen is repeated every 21 days. The response will be evaluated every 2 cycles in the first 36 weeks and every 4 cycles from week 36 till the end of treatment.
  Interventions: Drug: Sintilimab; Drug: Chidamide

INTERVENTIONS:
Drug: Sintilimab — 200mg intravenously on day 1, every 21 days for 1 cycle, 96 weeks for protocol treatment
Drug: Chidamide — 20mg po per week continuously

SUMMARY:
This is a multicenter prospective single arm phase II study. The purpose of this study is to evaluate the safety and efficiency of Sintilimab combined with Chidamide in the treatment of relapsed/refractory cutaneous T-cell lymphoma.

DETAILED DESCRIPTION:
This is a single-arm phase 2 study with fixed does of combined Sintilimab and Chidamide regimen. This regimen is repeated every 21 days. Sintilimab (200mg) is administered intravenously on day 1 of every cycle. Chidamide is used 20mg twice per week continuously. From the beginning of the trial, sindilimab will be used for 96 weeks, until disease progress, intolerable toxicity or patient/investigator discretion. Patients will continue to receive Chidamide treatment until disease progression, unacceptable toxicity, or patient/investigator discretion.

The response will be evaluated every 2 cycles in the first 36 weeks and every 4 cycles from week 36 till the end of treatment. The patients who achieve complete remission (CR), partial remission (PR), and stable disease (SD) will receive further treatment. The patients with progressed disease (PD) will be continue on the treatment and reassess after 4-8 weeks to rule out false progression. On confirmation of PD , patients will be withdrawn from the trial and receive salvage regimens.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed cutaneous T-cell lymphoma according World Health Organization (WHO) classification.
* ECOG≤2
* Patients with measurable lesions, with or without extra-dermal lesions, clinical stage of IIB-IVB.
* Patients received at least one systemic treatment previously and achieved no remission or relapsed after first-line treatment.
* Absolute neutrophil count (ANC）≥0.75×109/L，platelet (PLT) ≥ 50×109/L，hemoglobin (HGB）≥ 80 g/L
* Thyroid stimulating hormone (TSH) within normal range

Exclusion Criteria:

* Pre-existing uncontrolled active infection
* Alanine aminotransferase (ALT) >3 times upper limit of normal (ULN), total bilirubin (TBIL) >1.5 times ULN, serum creatinine >1.5 times ULN
* Patients with clinically significant QT interval prolongation (male > 450ms, female > 470ms), ventricular tachycardia (VT), atrial fibrillation (AF), acute coronary syndrome (ACS) within 1 year, congestive heart failure (CHF), and symptomatic coronary heart disease.
* Patients who have received organ transplantation or hematopoietic stem cell transplantation.
* Active bleeding or recent thrombotic disease
* Patients with known interstitial lung disease
* Patients with active autoimmune disease or history of autoimmune disease in the past 2 years
* Patients with CNS involvement
* Pregnant or lactating women
* History of mental illness

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | From date of signing the informed consent until the date of first confirmed progression or date of death from any cause, whichever came first, assessed up to 104 weeks
  ORR was defined as the proportion of patients who achieved CR or PR as their best response.

SECONDARY OUTCOMES:
Adverse Events | From date of signing the informed consent until the date of first confirmed progression or date of death from any cause, whichever came first, assessed up to 104 weeks
  Graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Duration of response (DOR) | From date of signing the informed consent until the date of first confirmed progression or date of death from any cause, whichever came first, assessed up to 104 weeks
  DOR was defined as the time from the first occurrence of CR or PR to the first diagnosis of PD or relapse.
Progression-Free Survival (PFS) | PFS was defined as interval from patient enrollment to the date of disease progression or death from any cause, whichever came first, assessed up to 104 weeks
  PFS was defined as interval from patient enrollment to the date of disease progression or death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No